CLINICAL TRIAL: NCT06685185
Title: A Study Investigating Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Doses of NNC0363-1063 in Healthy Participants and Participants With Type 1 Diabetes
Brief Title: A Research Study of a New Medicine NNC0363-1063 in Healthy Participants and Participants With Type 1 Diabetes
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN1644-7794; 2024-511808-17 (Other: European Medical Agency (EMA)); U1111-1304-2544 (Other: World Health Organization (WHO))
Record Dates: First submitted 2024-11-09; First posted 2024-11-12 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — insulin degludec; Insulin Detemir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part 1 SAD and Part 3 Meal test are double-blind study parts. Sponsor staff involved in the clinical trial is masked according to company standard procedures. Part 2 is open-label study part.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Part 1A: SAD: NNC0363-1063 (Experimental): Participants will receive single dose of NNC0363-1063 subcutaneously.
  Interventions: Drug: NNC0363-1063
- Part 1A: SAD: Placebo (Placebo Comparator): Participants will receive NNC0363-1063 matching placebo subcutaneously.
  Interventions: Drug: Placebo
- Part 1B: SAD: NNC0363-1063 (Experimental): Participants will receive NNC0363-1063 subcutaneously.
  Interventions: Drug: NNC0363-1063
- Part 1B: SAD: Insulin degludec (Active Comparator): Participants will receive insulin degludec subcutaneously.
  Interventions: Drug: Insulin degludec
- Part 2: PoP: NNC0363-1063 (Experimental): Participants will receive NNC0363-1063 subcutaneously.
  Interventions: Drug: NNC0363-1063
- Part 3 Meal test: NNC0363-1063 (Experimental): Participants will receive NNC0363-1063 subcutaneously.
  Interventions: Drug: NNC0363-1063
- Part 3 Meal test: Insulin detemir (Active Comparator): Participants will receive insulin detemir subcutaneously.
  Interventions: Drug: Insulin detemir

INTERVENTIONS:
Drug: NNC0363-1063 — NNC0363-1063 will be administered subcutaneously.
  Arms: Part 1A: SAD: NNC0363-1063; Part 1B: SAD: NNC0363-1063; Part 2: PoP: NNC0363-1063; Part 3 Meal test: NNC0363-1063
Drug: Placebo — Placebo will be administered subcutaneously.
  Arms: Part 1A: SAD: Placebo
Drug: Insulin degludec — Insulin degludec will be administered subcutaneously.
  Other Names: Tresiba
  Arms: Part 1B: SAD: Insulin degludec
Drug: Insulin detemir — Insulin detemir will be administered subcutaneously.
  Other Names: Levemir
  Arms: Part 3 Meal test: Insulin detemir

SUMMARY:
This study will look into testing a new medicine called NNC0363-1063 which may be used to treat people with diabetes. The study consists of three parts: Part 1 is a single ascending dose (SAD) study that comprises two subtypes: Part 1A conducted in healthy participants and Part 1B conducted in participants with type 1 diabetes (T1D). This study part will last for about 1½ to 5½ weeks. Part 2 is a proof-of-principle (PoP) study part conducted in participants with T1D and will last for about 3½ to 8½ weeks. Part 3 is a meal test multiple dose study part conducted in participants with T1D and will last for 7 to 11 weeks.

ELIGIBILITY:
Inclusion Criteria:

Part 1A SAD (healthy participants)

* Male or female of non-child bearing potential. Non-child bearing potential being defined as surgically sterilised (i.e. documented hysterectomy, bilateral salpingectomy or bilateral oophorectomy) or being postmenopausal (defined as no menses for 12 months without an alternative medical cause) prior to the day of screening.
* Age 18-64 years (both inclusive) at the time of signing the informed consent.
* Body mass index between 18.5-29.9 kilogram per square metre( kg/m^2) (both inclusive) at the day of screening.
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Part 1B SAD, Part 2 PoP and Part 3 Meal test (participants with T1D)

* Male or female of non-child bearing potential. Non-child bearing potential being defined as surgically sterilised (i.e. documented hysterectomy, bilateral salpingectomy or bilateral oophorectomy) or being postmenopausal (defined as no menses for 12 months without an alternative medical cause) prior to the day of screening.
* Age 18-64 years (both inclusive) at the time of signing the informed consent.
* Body mass index between 18.5-29.9 kg/m^2 (both inclusive) at the day of screening.
* Diagnosed with type 1 diabetes mellitus greater than or equal to( ≥)1 year prior to the day of screening.
* Considered to be generally healthy (except for mild conditions under stable treatment associated with type 1 diabetes mellitus) based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

Part 1A SAD (healthy participants)

* Male of reproductive age who, or whose female partner(s), is not using an adequate contraceptive method.
* Any condition, which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol.

Part 1B SAD, Part 2 PoP and Part 3 Meal test (participants with T1D)

* Male of reproductive age who, or whose female partner(s), is not using an adequate contraceptive method.
* Any condition, except for mild conditions under stable treatment associated with type 1 diabetes mellitus, which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 154 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Part 1 SAD: Number of adverse events | From investigational medicinal product (IMP) administration (day 1) until end of study visit (day 8)
  Measured in number of events.
Part 2 PoP: CL/F,I1063,SD- Apparent serum clearance of NNC0363-1063 after a single dose | From IMP administration at day 1 up to 7 days
  Measured in millilitre per hour*kilogram (mL/[h*kg]).
Part 3 Meal test: AUC,PG,meal: Area under the plasma glucose concentration-time curve at steady state | At day 2 of visit 2 and visit 3 after initiation of meal test
  Measured in hours*millimoles per litre (h*mmol/L).

SECONDARY OUTCOMES:
Part 1 SAD: Number of hypoglycaemic episodes | From investigational medicinal product (IMP) administration (day 1) until end of study visit (day 8)
  Measured in number of episodes.
Part 1 SAD: AUC0-inf,I1063,SD: Area under the serum NNC0363-1063 concentration-time curve from 0 to infinity after a single dose | Up to 7 days
  Measured in hours*picomoles per litre (h*pmol/L).
Part 1 SAD: AUC,I1063,SD- Area under the serum NNC0363-1063 concentration time curve after a single dose | Up to 2 days
  Measured in h*pmol/L.
Part 1 SAD: Cmax,I1063,SD- Maximum observed serum NNC0363-1063 concentration after a single dose | Up to 7 days
  Measured in picomoles per litre (pmol/L).
Part 2 PoP: AUC0-inf,I1063,SD: Area under the serum NNC0363-1063 concentration-time curve from 0 to infinity after a single dose | Up to 7 days
  Measured in h*pmol/L.
Part 2 PoP: AUC,I1063,SD- Area under the serum NNC0363-1063 concentration time curve after a single dose | Up to 2 days
  Measured in h*pmol/L.
Part 2 PoP: Cmax,I1063,SD- Maximum observed serum NNC0363-1063 concentration after a single dose | Up to 7 days
  Measured in pmol/L.
Part 3 Meal test: AUC0-1h,PG,meal: Area under the plasma glucose concentration-time curve from 0 to 1 hour after initiation of the meal test at steady state | From 0 hours to 1 hour after initiation of the meal test (day 2 of visit 2 and visit 3)
  Measured in h*mmol/L.
Part 3 Meal test: AUC0-2h,PG,meal: Area under the plasma glucose concentration-time curve from 0 to 2 hours after initiation of the meal test at steady state | From 0 hours to 2 hours after initiation of the meal test (day 2 of visit 2 and visit 3)
  Measured in h*mmol/L.
Part 3 Meal test: AUC0-4h,PG,mean: Area under the plasma glucose concentration-time curve from 0 to 4 hours after initiation of the meal test at steady state | From 0 hours to 4 hours after initiation of the meal test (day 2 of visit 2 and visit 3)
  Measured in h*mmol/L.
Part 3 Meal test: AUC0-6h,PG,meal: Area under the plasma glucose concentration-time curve from 0 to 6 hours after initiation of the meal test at steady state | From 0 hours to 6 hours after initiation of the meal test (day 2 of visit 2 and visit 3)
  Measured in h*mmol/L.
Part 3 Meal test: PGmax,meal: Maximum observed plasma glucose concentration at steady state | At day 2 of visit 2 and visit 3 after initiation of meal test
  Measured in millimoles per litre (mmol/L).
Part 3 Meal test: tPGmax,meal: Time to maximum observed plasma glucose concentration from at steady state | At day 2 of visit 2 and visit 3 after initiation of meal test
  Measured in hours.
Part 3 Meal test: ΔPGav,0-1h,meal: Mean change in plasma glucose from 0 to 1 hour after initiation of the meal test at steady state | From 0 hours to 1 hour after initiation of the meal test (day 2 of visit 2 and visit 3)
  Measured in mmol/L.
Part 3 Meal test: ΔPGav,0-2h,meal: Mean change in plasma glucose from 0 to 2 hours after initiation of the meal test at steady state | From 0 hours to 2 hours after initiation of the meal test (day 2 of visit 2 and visit 3)
  Measured in mmol/L.
Part 3 Meal test: AUCτ,I1063,SS: Area under the serum NNC0363-1063 concentration-time curve during one dosing interval at steady state | At day 2 of visit 2 and visit 3 after last IMP administration
  Measured in h*pmol/L.
Part 3 Meal test: Cmax,I1063,SS: Maximum observed serum NNC0363-1063 concentration during one dosing interval at steady state | At day 2 of visit 2 and visit 3 after last IMP administration
  Measured in pmol/L.
Part 3 Meal test: Number of adverse events | From first IMP administration (day 1 of visit 2 and visit 3) until 24 hours after last IMP administration (day 2 of visit 2 and visit 3)
  Measured in number of events.
Part 3 Meal test: Number of hypoglycaemic episodes | From first IMP administration (day 1 of visit 2 and visit 3) until 24 hours after last IMP administration (day 2 of visit 2 and visit 3)
  Measured in number of episodes.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com